CLINICAL TRIAL: NCT01485718
Title: Effect of Daily Glucomannan in Overweight Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: ProMedica Health System (Other)
Responsible Party: Principal Investigator, Katherine Cochran, PGY1-Pharmacy Resident, ProMedica Health System
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11-117
Record Dates: First submitted 2011-11-26; First posted 2011-12-05 (Estimated); Last update posted 2011-12-13 (Estimated); Status verified 2011-12

CONDITIONS: Overweight; Obesity
Keywords: Obesity; Overweight; Weight loss
MeSH Terms: conditions — Overweight; Obesity; Weight Loss | interventions — (1-6)-alpha-glucomannan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glucomannan (Active Comparator): Participants in the glucomannan arm will receive glucomannan 2 capsules 30 minutes before the three largest meals of the day.
  Interventions: Dietary Supplement: Glucomannan
- Placebo (Placebo Comparator): Participants in the placebo arm will receive placebo 2 capsules 30 minutes before the three largest meals of the day.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Glucomannan — Participants in the glucomannan arm will receive glucomannan 2 capsules 30 minutes before the three largest meals of the day for 12 weeks
  Arms: Glucomannan
Dietary Supplement: Placebo — Participants in the placebo arm will receive placebo 2 capsules 30 minutes before the three largest meals of the day.
  Arms: Placebo

SUMMARY:
Glucomannan is a dietary supplement that has been marketed for weight loss. There is some research that supports this claim but more research is necessary. This is research study is being conducted to determine if the dietary supplement glucomannan is effective for weight loss in adults greater than 18 years of age who are overweight.

Participants will be randomized in a 1:1 manner (like the flip of a coin) to receive either glucomannan 575 milligrams, 2 capsules three times daily or placebo, 2 capsules three times daily. The study will last for 12 weeks.

At the start of the study participants will be asked questions about current medications and diet/exercise regimen, a weight and height will be obtained, and they will be given a one-month's supply of study supplement. An investigator will call each participant after they have been taking the supplement for 2 weeks to ensure that the participant is tolerating the supplement and answer any questions. Throughout the study, participants will be required to follow-up with investigators in the office every 4 weeks (a total of 3 follow-up appointments). Every 4 weeks, the investigators will weigh participants, count the leftover capsules from the previous month, and ask about any adverse effects you may be experiencing. At the conclusion of the study, a final weight will be compared with the baseline weight to determine if the medication had an effect on weight loss.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years old
* Overweight (BMI ≥ 25 kg/m2)

Exclusion Criteria:

* Pregnant or nursing women
* Women of childbearing age will be excluded unless they are on some form of contraception
* Participation in any other formal or informal weight reduction program

  1. Currently enrolled in another weight loss study
  2. Currently enrolled in a weight loss program
  3. Active attempt to lose weight with diet and/or exercise within the last month
  4. Currently on one of the following medications known to cause weight loss:

     * Alli/Xenical(orlistat)
     * Adipex-P (phentermine)
     * Bontril (phendimetrazine)
     * Dexoxyn (methamphetamine)
     * Didrex (benzphetamine)
     * Tenuate (diethylpropion)
     * Meridia (sibutramine)
     * Byetta (exenatide) or Victoza (liraglutide)
     * Stimulants
* Recently (within the last three months) started on any medication that may cause weight gain
* A diagnosis of heart failure
* Structural abnormalities of the esophagus or gut
* Previous GI surgery for weight reduction
* Inflammatory bowel or irritable bowel disease
* A life expectancy of <6 months
* Allergy to glucomannan or any component of the placebo

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-10; Primary Completion 2012-03 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Weight | 12 weeks
  The primary outcome is the difference between weight at 12 weeks and the baseline weight.

SECONDARY OUTCOMES:
Side Effects | Assessed at 2, 4, 8, and 12 week intervals
  Patient reported side effects assessed at each patient visit. Specifically side effects related to gastrointestinal function.

CONTACTS AND LOCATIONS:
Overall Officials: Steve Smith, MS, RPh, Study Director — The Toledo Hospital; Ashley M Parrott, PharmD, Study Chair — The Toledo Hospital; Louito Edje, MD, Study Chair — The Toledo Hospital; Lindsey Bostelman, MD, Study Chair — The Toledo Hospital; David Knieriem, Study Chair — The Toledo Hospital
Locations (1):
- W.W. Knight Family Practice Center, Toledo, Ohio, United States